CLINICAL TRIAL: NCT06158126
Title: UNCPM 22314 - Evaluating the Safety of Pregnancy, Infant and Maternal Health Outcomes Among PrEP Users in Malawi
Brief Title: UNCPM 22314 - Pregnancy, Infant and Maternal Health Outcomes Study
Acronym: PrIMO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); United States President's Emergency Plan for AIDS Relief (U.S. Federal Agency); Ministry of Health, Malawi (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-2220; 1P01HD112215 (NIH)
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Pre-exposure Prophylaxis; HIV Prevention; Pregnancy Related
Keywords: PrEP; Pregnancy; Breastfeeding; Infant health; HIV prevention; Maternal health; Eliminating mother-to-child transmission (EMTCT)
MeSH Terms: conditions — Breast Feeding | interventions — Tenofovir; Racivir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral PrEP (FTC/TDF or TDF/3TC) during pregnancy (Active Comparator): The arm will include pregnant women who have met eligibility criteria, consented, and chosen to initiate or remain on oral PrEP (FTC/TDF or TDF/3TC) during pregnancy. Within the arm, they will be grouped according to whether they started oral PrEP before or after pregnancy diagnosis. All participants will continue to be offered oral PrEP throughout the study and will be followed up for the duration of the study. All women will be registered into the PrEP Pregnancy Registry as part of routine care.
  Interventions: Drug: Initiating daily oral PrEP during pregnancy; Drug: Already using daily oral PrEP at the time of pregnancy diagnosis
- Long-acting injectable cabotegravir (CAB-LA) during pregnancy (Experimental): The arm will include pregnant women who have met eligibility criteria, consented, and chosen to initiate or remain on injectable PrEP (CAB-LA) during pregnancy. Within the arm, they will be grouped according to whether they started CAB-LA before or after pregnancy diagnosis. All participants will continue to be offered CAB-LA throughout the study and will be followed up for the duration of the study. All women will be registered into the PrEP Pregnancy Registry as part of routine care.
  Interventions: Drug: Initiating injectable PrEP during pregnancy; Drug: Already using injectable PrEP (CAB-LA) at the time of pregnancy diagnosis

INTERVENTIONS:
Drug: Initiating daily oral PrEP during pregnancy — Group 1a will include pregnant women who initiate oral PrEP when already pregnant, at enrollment into the study.
  Other Names: Tenofovir disoproxil fumarate (TDF)/emtricitabine (FTC) or lamivudine (3TC) (FTC/TDF or TDF/3TC)
  Arms: Oral PrEP (FTC/TDF or TDF/3TC) during pregnancy
Drug: Already using daily oral PrEP at the time of pregnancy diagnosis — Group 1b will include women already using daily oral PrEP at the time of pregnancy diagnosis and enrollment in the study.
  Other Names: Tenofovir disoproxil fumarate (TDF)/emtricitabine (FTC) or lamivudine (3TC) (FTC/TDF or TDF/3TC)
  Arms: Oral PrEP (FTC/TDF or TDF/3TC) during pregnancy
Drug: Initiating injectable PrEP during pregnancy — Group 2a will include pregnant women who initiate injectable PrEP (CAB-LA) when already pregnant, at enrollment into the study.
  Other Names: CAB-LA
  Arms: Long-acting injectable cabotegravir (CAB-LA) during pregnancy
Drug: Already using injectable PrEP (CAB-LA) at the time of pregnancy diagnosis — Group 2b will include women using injectable PrEP (CAB-LA) at the time of pregnancy diagnosis and enrollment into the study.
  Other Names: CAB-LA
  Arms: Long-acting injectable cabotegravir (CAB-LA) during pregnancy

SUMMARY:
The primary purpose of this study is to assess the safety of long-acting injectable cabotegravir (CAB-LA) and oral pre-expose prophylaxis (PrEP) (FTC/TDF or 3TC/TDF) for the prevention of HIV during pregnancy and breastfeeding among pregnant women and their infants in Malawi. The main question the study aims to answer is:

- Do composite adverse pregnancy events, maternal health outcomes, and/or infant health outcomes differ between individuals taking oral PrEP and those taking CAB-LA?

Women who are already using PrEP at the time of pregnancy diagnosis or those who initiate PrEP during pregnancy will enroll into a Safety Cohort where they will be closely followed up during pregnancy while optimizing their antenatal care (ANC) per the Malawi ANC package. Women will have access to either CAB-LA or oral PrEP and will be given an opportunity to choose one option. Women and their infants will attend a series of follow-up visits through pregnancy, birth, and the postnatal period.

In addition, the study will contribute to the development of a national PrEP Pregnancy Registry which will be initially rolled out in Lilongwe and Blantyre -the two most populous cities in Malawi-before a nationwide roll out begins under the guidance of the Malawi Ministry of Health.

DETAILED DESCRIPTION:
For the prospective safety cohort, the study will enroll and follow up eligible women attending antenatal clinic and planning to deliver at Bwaila District Hospital in Lilongwe, Malawi. The primary objective is comparing composite adverse pregnancy events (spontaneous miscarriage, stillbirth, preterm birth, or infant born small for gestational age) between women using CAB-LA and those using oral PrEP. Pregnant women assessed as being at substantial risk for HIV and eligible for PrEP per Malawi national guidelines will be included. Infants will be followed alongside their mothers.

All women meeting eligibility criteria will be consented and offered PrEP (if not already taking it). Women will have access to either CAB-LA or oral PrEP and will be given an opportunity to choose one option. For the Safety Cohort, researchers will group women according to use of oral PrEP (FTC/TDF or TDF/3TC) versus injectable PrEP (CAB-LA), and according to PrEP use before or after pregnancy diagnosis as follows:

Group 1a: Initiating daily oral PrEP during pregnancy Group 1b: Using daily oral PrEP at the time of pregnancy diagnosis Group 2a: Initiating injectable CAB-LA during pregnancy Group 2b: Using injectable CAB-LA at the time of pregnancy diagnosis.

Follow-up contacts for the mother-infant pairs will follow the Malawi ANC package schedule of events during pregnancy, and then include a delivery/birth visit and a series of postpartum visits through week 52 (exit visit). Interim visits initiated by the study could be to repeat abnormal laboratory tests or for safety monitoring of an adverse event. Interim visits initiated by the participant could be to report an adverse event or to seek primary care. Visits will include a series of clinical and laboratory procedures to monitor and assess any pregnancy, maternal health, or infant adverse outcomes. All clinical and laboratory adverse events will be accessed and graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events. These follow up visits will also optimize antenatal care per the Malawi ANC package.

Clinical and sociodemographic data with be collected by the clinic staff at the UNC study site at Bwaila District Hospital. Quantitative methods will involve administration of brief behavioral surveys conducted every six months during the study follow up period. The surveys will include (but not be limited to) questions about women's attitudes and beliefs about the two PrEP options, and questions about product-related choice and preferences. Surveys will also include risk questionnaire collecting information about previous sexual activity, partners, and PrEP use over the preceding six months, as well as self-perception of HIV risk.

As part of the mixed methods approach, researchers will also conduct qualitative interviews with women to further assess acceptability of oral PrEP or CAB-LA at enrollment, 6 weeks postnatal, and study exit. This component will include a series of in-depth interviews (IDIs) with a subset of women from each group, as well as IDIs with a subset of women who experience adverse obstetric outcomes and those who seroconvert while on injectable or oral PrEP. The aim is to assess whether there are changes in the perceptions and acceptability of oral PrEP or CAB-LA over the study period and explore women's views about future PrEP use during pregnancy and breastfeeding and their choices to use PrEP with subsequent pregnancies.

Additionally, all women in the safety cohort will be enrolled into a PrEP in Pregnancy Registry. The registry in this study will contribute to the development of a national PrEP Pregnancy Registry and subsequent registration and longitudinal surveillance of eligible women without HIV at CAB-LA early access sites in Blantyre and Lilongwe. The registry will include all women initiating PrEP in the national program while pregnant or at the time of diagnosis of pregnancy, and those who become pregnant while on PrEP.

Registry administrators (RAs) at PrEP sites, who may be community health workers, nurses or midwives working at these sites, will register pregnant women into the PrEP Pregnancy Registry as part of routine data collection. The RA's will then obtain basic health information at enrollment, and conduct a follow-up visit at or following delivery to collect pregnancy outcomes and health care provided during delivery. These activities will be conducted as part of routine care.

ELIGIBILITY:
Inclusion Criteria:

Maternal participants:

* Confirmed pregnancy by urine pregnancy test or ultrasound.
* Aged 15 years or older
* PrEP-eligible by Malawi local guidelines
* Confirmed HIV-negative based on the local HIV testing algorithm
* Hepatitis B surface antigen (HBsAg) negative
* Weight >35 kg
* Provided informed consent and expressed willingness to participate in study activities with their infants.

Infant participants: Infant participants will enter the study with their mother as unborn infants. There are no specific eligibility criteria for infant participation otherwise.

Exclusion Criteria:

Maternal participants will not be eligible to enter the prospective cohort study if any of the following conditions are identified during the screening process:

* Known to be living with HIV
* Known allergies to CAB-LA, TDF/3TC or FTC/TDF
* Other current significant disease process (active or chronic), substance use, or social circumstances that, in the judgment of the site investigator would make participation in the study unsafe.
* Intention to leave the study site's catchment area of Bwaila before scheduled study exit.

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women
Enrollment: 621 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of composite adverse pregnancy outcomes | Enrollment through birth
  Rate will be calculated as the number of women with an adverse pregnancy outcome, defined as the occurrence of any one of the following events: spontaneous miscarriage (pregnancy lost before 28 weeks gestation), stillbirth (fetal death at or after 28 weeks gestation), preterm birth (delivery before 37 weeks gestation), infant born small for gestational age (birth weight of less than 10th percentile for gestational age) over the accumulated person time from enrollment through birth.

SECONDARY OUTCOMES:
Proportion of women developing grade 3 or higher clinical or laboratory events | Enrollment through 52 weeks postpartum
  Proportions will be calculated as the number of women developing grade three or higher clinical or laboratory events over the total number of enrollees in the cohort. Grade 3 or higher clinical or laboratory events will be assessed and graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Proportion of infants developing stage 3 or higher clinical or laboratory events | Birth through 52 weeks of life
  Proportions will be calculated as the number of infants developing stage three or higher clinical or laboratory events over the total number of infants in the cohort. Stage 3 or higher clinical or laboratory events will be accessed and graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Proportion of infants born with congenital anomalies | Birth through 52 weeks of life
  Proportions will be calculated as the number of infants born with congenital anomalies over the total number of infants in the cohort. Congenital anomalies will be diagnosed with neonatal surface exam and fetal anatomic ultrasound
Number of infants who are underweight | Birth through 52 weeks of life
  Number of infants who are underweight, defined as weight for age z-score (WAZ) <-2, assessed at weeks 1, 6, 12, 26 and 52 weeks after birth.
Proportion of infants who are underweight | Birth through 52 weeks of life
  Proportions will be calculated as the number of infants who are underweight over the total number of infants in the cohort. Underweight will be defined as weight for age z-score (WAZ) <-2, assessed at weeks 1, 6, 12, 26 and 52 weeks after birth.
Number of infants who are stunted | Birth through 52 weeks of life
  A child will be considered stunted if s/he has a length for age z-score (LAZ) <-2, assessed at weeks 1, 6, 12, 26 and 52 after birth.
Proportion of infants who are stunted | Birth through 52 weeks of life
  Proportions will be calculated as the number of infants who are stunted over the total number of infants in the cohort. Infants will be considered stunted if s/he has a length for age z-score (LAZ) <-2, assessed at weeks 1, 6, 12, 26 and 52 after birth.
Number of infants who have moderate or severe acute malnutrition | Birth through 52 weeks of life
  Malnourishment based on anthropometrics per World Health Organization (WHO) definitions. Moderate acute malnutrition defined as a weight for length z-score (WLZ) between -3 and <-2, or mid-upper arm circumference (MUAC) between 115 millimeters and <125 millimeters. Severe acute malnutrition defined as a weight for length z-score (WLZ) of < -3 or MUAC < 115 millimeters, or the presence of bilateral pitting edema, or both. Assessed at weeks 1, 6, 12, 26 and 52 after birth.
Proportion of infants who have moderate or severe acute malnutrition | Birth through 52 weeks of life
  Proportions will be calculated as the number of infants who have moderate or severe acute malnutrition over the total number of infants in the cohort. Malnourishment based on anthropometrics per World Health Organization (WHO) definitions. Moderate acute malnutrition defined as a weight for length z-score (WLZ) between -3 and <-2, or mid-upper arm circumference (MUAC) between 115 millimeters and <125 millimeters. Severe acute malnutrition defined as a weight for length z-score (WLZ) of < -3 or MUAC < 115 millimeters, or the presence of bilateral pitting edema, or both. Assessed at weeks 1, 6, 12, 26 and 52 after birth.
Number of infants with poor neurodevelopment outcomes | Birth through 52 weeks of life
  Defined as a low Caregiver-Reported Early Development Index (CREDI) and/or Mullen Scales of Early Learning (MSEL) score for age, assessed at weeks 1, 6, 12, 26 and 52 after birth
Acceptability of oral PrEP or CAB-LA | Delivery through 52 weeks postpartum
  Based on analysis of in-depth interviews with approximately 50 women in the study. Content analysis and NVivo version 1.7 will be used to develop a codebook using domains and constructs from theoretical framework for acceptability by Sekhon. Data will then be displaced on matrices using the framework to display the patterns emerging from the text. Assessed at delivery, 12 weeks postpartum, and 52 weeks postpartum
Adoption of PrEP in Pregnancy Registry | 6 to 24 months after implementation
  Adoption will be defined as the number of targeted settings (including districts, sites, and providers) who initiated register use by the end of the study. Adoption will be assessed at 6, 12, and 24 months after register implementation.
Reach of PrEP in Pregnancy Registry | 6 to 24 months after implementation
  Reach will be defined as the total number of entries in the register at each site. Reach will be assessed at 6, 12, and 24 months after register implementation.
Fidelity to PrEP in Pregnancy Registry | 6 to 24 months after implementation
  Fidelity is defined as the number of pregnant women who have complete entries for all infant and obstetric outcomes in the register as per protocol. Fidelity will be assessed at 6, 12, and 24 months after register implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Friday Saidi, MBBS, MMED, Principal Investigator — UNC Project Malawi
Locations (1):
- Bwaila Distict Hospital, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC
URL: http://unc.edu

REFERENCES:
- [Derived] Saidi F, Shah S, Squibb M, Chinula L, Nakanga C, Mvalo T, Matoga M, Bula AK, Chagomerana MB, Kamanga F, Kumwenda W, Mkochi T, Masiye G, Moya I, Herce ME, Rutstein SE, Thonyiwa V, Nyirenda RK, Mwapasa V, Hoffman I, Hosseinipour MC. Evaluating the impact of HIV pre-exposure prophylaxis on pregnancy, infant, and maternal health outcomes in Malawi: PrIMO study protocol. BMC Public Health. 2024 Sep 27;24(1):2604. doi: 10.1186/s12889-024-20029-3. PMID 39334032